CLINICAL TRIAL: NCT01135576
Title: Iron Fortified Beverages and Application in Women Predisposed to Anemia
Acronym: FeDrink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Grupo Leche Pascual (Unknown); Madrid Salud, Madrid, Spain (Unknown)
Responsible Party: Principal Investigator, M Pilar Vaquero, Scientific Researcher, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGL2006/09519/ALI
Record Dates: First submitted 2010-05-28; First posted 2010-06-03 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Iron-deficiency Anemia
Keywords: Ferric pyrophosphate; Fortification; Fruit juice; Functional food; Bioavailability; iron status; Women; iron-deficiency anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo juices (Placebo Comparator): Consumption of non-iron fortified fruit juices as part of the usual diet
  Interventions: Dietary Supplement: non-fortified fruit juices consumed as part of the usual diet
- Iron fortified fruit juices (Experimental): Consumption of iron fortified fruit juices as part of the usual diet
  Interventions: Dietary Supplement: Iron fortified fruit juice

INTERVENTIONS:
Dietary Supplement: non-fortified fruit juices consumed as part of the usual diet
  Arms: Placebo juices
Dietary Supplement: Iron fortified fruit juice — Consumption of micronized iron pyrophosphate supplemented fruit juices as part of the usual diet
  Arms: Iron fortified fruit juices

SUMMARY:
* The objective of the study is to know if consumption of an iron fortified fruit juice containing micronized iron pyrophosphate, is useful to increase iron status in women predisposed to iron deficiency anemia.
* A secondary objective is to know if consumption of this iron fortified fruit juice modifies bone remodelling.

ELIGIBILITY:
Inclusion Criteria:

* Women
* non-smoker
* non-pregnant
* non-breastfeeding
* serum ferritin <40 ng/ml
* hemoglobin>=11g/dl

Exclusion Criteria:

* Serum Ferritin >=40 ng/ml
* Hemoglobin <11g/dl
* Amenorrhea
* Menopause
* Iron deficiency anemia
* Thalassemia
* Hemochromatosis
* Blood donors
* Chronic gastric diseases
* Renal diseases
* Eating disorders
* Allergy to any component of the study juices
* Consumption of iron or ascorbic acid supplements within 4 month prior to participating in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Serum Ferritin | monitored during 16 weeks

SECONDARY OUTCOMES:
Serum transferrin | monitored during 16 weeks
Hemoglobin | monitored during 16 weeks
serum iron | monitored during 16 weeks
transferrin saturation | monitored during 16 weeks
soluble transferrin receptor | monitored during 16 weeks
zinc protoporphyrin | monitored during 16 weeks
Total red blood cells | monitored during 16 weeks
Hematocrit | monitored during 16 weeks
Mean corpuscular volume | monitored during 16 weeks
Red blood cell distribution width | monitored during 16 weeks
25-hydroxycholecalciferol | monitored during 16 weeks
alkaline phosphatase bone-isoenzyme (ALP) | monitored during 16 weeks
serum cross-linked N-telopeptide of type I collagen (NTx) | monitored during 16 weeks
Total cholesterol | monitored during 16 weeks
HDL-cholesterol | monitored during 16 weeks
LDL-cholesterol | monitored during 16 weeks
Glucose | monitored during 16 weeks
Serum triacylglycerols | monitored during 16 weeks
T-chol/HDL-chol | monitored during 16 weeks
LDL-chol/HDL-chol | monitored during 16 weeks
Systolic blood pressure | monitored during 16 weeks
Diastolic blood pressure | monitored during 16 weeks

REFERENCES:
- [Background] Navas-Carretero S, Perez-Granados AM, Schoppen S, Sarria B, Carbajal A, Vaquero MP. Iron status biomarkers in iron deficient women consuming oily fish versus red meat diet. J Physiol Biochem. 2009 Jun;65(2):165-74. doi: 10.1007/BF03179067. PMID 19886395
- [Background] Navas-Carretero S, Perez-Granados AM, Schoppen S, Vaquero MP. An oily fish diet increases insulin sensitivity compared to a red meat diet in young iron-deficient women. Br J Nutr. 2009 Aug;102(4):546-53. doi: 10.1017/S0007114509220794. Epub 2009 Feb 12. PMID 19210857
- [Background] Navas-Carretero S, Perez-Granados AM, Sarria B, Vaquero MP. Iron absorption from meat pate fortified with ferric pyrophosphate in iron-deficient women. Nutrition. 2009 Jan;25(1):20-4. doi: 10.1016/j.nut.2008.07.002. Epub 2008 Aug 26. PMID 18752926
- [Background] Navas-Carretero S, Perez-Granados AM, Sarria B, Carbajal A, Pedrosa MM, Roe MA, Fairweather-Tait SJ, Vaquero MP. Oily fish increases iron bioavailability of a phytate rich meal in young iron deficient women. J Am Coll Nutr. 2008 Feb;27(1):96-101. doi: 10.1080/07315724.2008.10719680. PMID 18460487
- [Background] Navas-Carretero S, Sarria B, Perez-Granados AM, Schoppen S, Izquierdo-Pulido M, Vaquero MP. A comparative study of iron bioavailability from cocoa supplemented with ferric pyrophosphate or ferrous fumarate in rats. Ann Nutr Metab. 2007;51(3):204-7. doi: 10.1159/000104138. Epub 2007 Jun 18. PMID 17587790
- [Background] Sarria B, Navas-Carretero S, Lopez-Parra AM, Perez-Granados AM, Arroyo-Pardo E, Roe MA, Teucher B, Vaquero MP, Fairweather-Tait SJ. The G277S transferrin mutation does not affect iron absorption in iron deficient women. Eur J Nutr. 2007 Feb;46(1):57-60. doi: 10.1007/s00394-006-0631-x. Epub 2007 Jan 5. PMID 17206377
- [Background] Navas-Carretero S, Pérez-Granados AM, Sarriá B, Schoppen S, Vaquero MP. Iron bioavailability from pate enriched with encapsulated ferric pyrophosphate or ferrous gluconate in rats. Food Sci Tech Int 13:159-163, 2007.
- [Background] Toxqui L, De Piero A, Courtois V, Bastida S, Sanchez-Muniz FJ, Vaquero MP. [Iron deficiency and overload. Implications in oxidative stress and cardiovascular health]. Nutr Hosp. 2010 May-Jun;25(3):350-65. Spanish. PMID 20593115
- [Result] Blanco-Rojo R, Perez-Granados AM, Toxqui L, Zazo P, de la Piedra C, Vaquero MP. Relationship between vitamin D deficiency, bone remodelling and iron status in iron-deficient young women consuming an iron-fortified food. Eur J Nutr. 2013 Mar;52(2):695-703. doi: 10.1007/s00394-012-0375-8. Epub 2012 May 23. PMID 22618893
- [Result] Blanco-Rojo R, Perez-Granados AM, Toxqui L, Gonzalez-Vizcayno C, Delgado MA, Vaquero MP. Efficacy of a microencapsulated iron pyrophosphate-fortified fruit juice: a randomised, double-blind, placebo-controlled study in Spanish iron-deficient women. Br J Nutr. 2011 Jun;105(11):1652-9. doi: 10.1017/S0007114510005490. Epub 2011 Feb 8. PMID 21303569